CLINICAL TRIAL: NCT03640156
Title: To Mirror or Not to Mirror Upon Perceived Eye Contact? The Effect of Oxytocin on Socially Adaptive Mirror System Functioning in Autism
Brief Title: Modulating Socially Adaptive Mirror System Functioning in Autism by Oxytocin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Alaerts, Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: S56327c
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Oxytocin; Eye Contact; Mirror System; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (OXT) spray (Experimental): Syntocinon nasal spray (product code RVG 03716) will be used to intranasally administer one single dose (24 IU) of OXT (3 puffs of 4 IU per nostril).
  Interventions: Drug: Oxytocin
- Placebo (PL) spray (Placebo Comparator): Physiological water (a solution of sodium chloride (NaCl) in water) will be used to intranasally administer one single dose (24 IU) of PL (3 puffs of 4 IU per nostril).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin — A single dose (24IU) of nasal spray (3 puffs of 4IU per nostril) will be administered before the assessment of the neurophysiological measures.
  Other Names: Syntocinon (product code RVG 03716)
  Arms: Oxytocin (OXT) spray
Other: Placebo — A single dose (24IU) of nasal spray (3 puffs of 4IU per nostril) will be administered before the assessment of the neurophysiological measures.
  Arms: Placebo (PL) spray

SUMMARY:
This study investigates the efficacy of a single-dose of exogenous oxytocin administration on socially adaptive mirror-motor mapping in participants with Autism Spectrum Disorders. A placebo-controlled cross-over trial will be conducted: each participant will receive both a single-dose of placebo and oxytocin in two sessions separated by one week. The order of nasal spray will be randomised across participants. Mirror-motor mapping will be assessed by transcranial magnetic stimulation (TMS), a standard technique to investigate mirror system activity.

DETAILED DESCRIPTION:
The brain's action observation network or 'mirror system' supports a variety of socio-cognitive functions, as it enables us to internally simulate and understand others' actions, emotions and intentions. Generally, mirror responses are larger upon the observation of actions accompanied by relevant information for the observer, such as direct eye contact from the actor. In other words, 'mirroring' is adaptively modulated according to the social salience of the observed actions (i.e. it is socially adaptive).

Individuals with Autism Spectrum Disorders (ASD) are known to endure difficulties with correctly recognizing eye contact as a communicative cue. Instead, they tend to experience eye contact as stressful and arousing. It is therefore hypothesized that, upon the observation of actions combined with salient gaze cues from the actor, these mirroring processes will not be adaptively modulated in participants with ASD.

As appropriate processing of eye contact is a key aspect of (non-verbal) communicative behavior, the investigator will investigate the efficacy of a single dose of intranasal oxytocin administration for enhancing socially-adaptive mirroring in ASD. Oxytocin is a neuropeptide that acts as a regulator social brain areas. On a behavioral level, it is known to enhance the saliency of observed social cues and to improve prosocial behavior. As such, it is regarded a promising intervention for alleviating the social and communicative deficits in ASD.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Young adults (between 18 - 35 y/o)
* Right-handed
* Official diagnosis of Autism Spectrum Disorders (for ASD participants)

Exclusion Criteria:

* Female
* Left-handed
* Any neuro(psycho)logical / psychiatric illness (for healthy controls)
* Motor dysfunctions of the hands / arms
* Any contradiction to TMS research as assessed with the TMS screening list: no metal objects in the body (e.g. pacemaker, coronary bypass clips, implants, medication pumps, ...), history of brain trauma in the past (e.g. meningitis, epilepsy, surgery, ...) or history of drug and/or alcohol abuse.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in socially adaptive mirroring as measured by TMS | 30 minutes after spray administration
  After a single dose of nasal spray, TMS will be applied to assess mirror-motor mapping during the observation of socially relevant vs. irrelevant visuomotor information.

SECONDARY OUTCOMES:
Change from baseline in mirroring of others' actions as measured by TMS | 30 minutes after spray administration
  After a single dose of nasal spray, TMS will be applied to assess basic mirror-motor mapping of observed actions.
Change from baseline in corticospinal excitability as measured by TMS | 30 minutes after spray administration
  After a single dose of nasal spray, TMS will be applied to assess corticospinal excitability when the participant is at rest (without any visuomotor information).
Change from baseline in total fixation duration towards the eye region of the model. | 30 minutes after spray administration
  During movement observation, participants' viewing behavior will be monitored by means of head-mounted eye tracking technology.

OTHER OUTCOMES:
Change from baseline in saliva-based oxytocin concentrations | Before and 60 minutes after spray administration
  Saliva samples will be collected before nasal spray administration and after the experimental procedure to be able to monitor the pharmacokinetics of oxytocin.
Change from baseline in Public Self-Awareness Score on Situational Self-Awareness Scale (SSAS) | 60 minutes after spray administration
  Informant-based self-report scale to assess public self-awareness in a specific situation as measured by SSAS. Likert scale: I totally agree (1) - I totally disagree (10); lower scores indicate more public self-awareness.
Change from baseline in Arousal and Pleasure on the Self-Assessment Manikin (SAM) | 60 minutes after spray administration
  Informant-based scale to assess self-reported arousal and pleasure in a specific situation as measured by SAM. Likert scale: Pleasant / Not aroused (1) - Unpleasant / Aroused (9). Higher scores indicate more arousal and less pleasure.

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Alaerts, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prinsen J, Bernaerts S, Wang Y, de Beukelaar TT, Cuypers K, Swinnen SP, Alaerts K. Direct eye contact enhances mirroring of others' movements: A transcranial magnetic stimulation study. Neuropsychologia. 2017 Jan 27;95:111-118. doi: 10.1016/j.neuropsychologia.2016.12.011. Epub 2016 Dec 8. PMID 27939365
- [Background] Prinsen J, Brams S, Alaerts K. To mirror or not to mirror upon mutual gaze, oxytocin can pave the way: A cross-over randomized placebo-controlled trial. Psychoneuroendocrinology. 2018 Apr;90:148-156. doi: 10.1016/j.psyneuen.2018.02.016. Epub 2018 Feb 22. PMID 29494953
- See also: Related Information — https://gbiomed.kuleuven.be/english/research/50000743/nrrg1/neuromodulation-laboratory